CLINICAL TRIAL: NCT03855930
Title: Phantom Limb Pain Triggered by Micturition, An Functional Magnetic Resonance Imaging (FMRI) Study in Lower Limb Amputees
Brief Title: Phantom Limb Pain Triggered by Micturition
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Loewenstein Hospital (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: 0012-18-LOE
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-01

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- micturition induced PLP: 10 Patients with chronic post amputation micturition induced PLP.All subjects must fulfill all of the inclusion criteria and meet none of the exclusion criteria.
  All patients will go through functional MRI study
  Interventions: Diagnostic Test: functional MRI
- non micturition induced PLP: 10 Patients with chronic post amputation with PLP and without post amputation micturition induced PLP All subjects must fulfill all of the inclusion criteria and meet none of the exclusion criteria.All patients will go through functional MRI study
  Interventions: Diagnostic Test: functional MRI
- healthy volunteers: 10 healthy volunteers. All patients will go through functional MRI study
  Interventions: Diagnostic Test: functional MRI

INTERVENTIONS:
Diagnostic Test: functional MRI — During the study, standard motor and sensory paradigms will be performed to establish anatomical and functional patterns in the non-painful state. The patient will then be asked to urinate (to an external collecting tube system).

SUMMARY:
Phantom Limb Pain ( PLP) is pain that is perceived and referred to a region of the body that is no longer present. in most patients, severity and frequency of phantom pain attacks gradually decrease over several weeks to 2 years following amputation, however in 5-10% significant pain remains a serious problem.

It has been hypothesized, that deprivation of various inputs from the limbs to the brain cause an abnormal neuro-signature to be produced generating cortical maladaptive neuroplasticity and reorganization. Areas representing the amputated body part are taken over by neighboring representational zones in both the somatosensory and motor cortex generating pain in absence of stimuli.

A seminal paper published by Lotze et al "Phantom movements and pain: a functional magnetic resonance imaging (fMRI) study in upper limb amputees. - participants had to pucker their lips at a metronome-paced speed while functional magnetic resonance images were taken. Only in amputees with phantom-limb pain did a shift of the mouth representation into the hand representation occur; those without pain and the healthy control do not display a similar shift.

Scarce reports have been made on a similar phenomenon- micturition induced lower limb phantom pain.

We speculate that a similar maladaptive central nerve system (CNS) plasticity in which this genital representation would invade cortical areas with somatotopic affiliation to the lower extremity could be implicated in the pathophysiology of this phenomenon.

DETAILED DESCRIPTION:
The present study was there for devised to examine this hypothesis utilizing fMRI imaging of temporo-spatial cortical activation during micturition and pain generation.

We hypothesis that in amputees with phantom-limb pain a shift of the genital representation into the leg representation will occur; and will be demonstrated as an uni-hemispheral activity on fMRI during micturition and pain suggesting maladaptive CNS plasticity. Moreover, we speculate that healthy volunteers will not display a similar shift.

During the study, standard motor and sensory paradigms will be performed to establish anatomical and functional patterns in the non-painful state. The patient will then be asked to urinate (to an external collecting tube system).

All anatomical data will be examined by a certified clinical imaging specialist to exclude concomitant brain pathology.

Study population -

1. 10 Patients with chronic post amputation micturition induced PLP.All subjects must fulfill all of the inclusion criteria and meet none of the exclusion criteria.
2. 10 Patients with chronic post amputation with PLP and without post amputation micturition induced PLP All subjects must fulfill all of the inclusion criteria and meet none of the exclusion criteria.
3. 10 healthy volunteers

FMRI data analysis signifying, statistically significant uni-spatial voxel activity during micturition, in the study group

ELIGIBILITY:
Inclusion Criteria:

* 9 months or more post amputation, no anatomical stump pathology
* Ambulatory and to comply with study protocol
* Suffering from significant pain (VAS>??). pain level has plateaued for at lest 2 months prior to enrolment.
* Pain is perceived to be located in the missing limb
* Pain level is brought up or increases (by at least 3 VAS points) by micturition.
* Maneuvers causing abdominal pressure elevation do not generate similar symptoms.
* Subject received an explanation about the nature of the study and agrees to provide written informed consent
* Subject is capable and willing to follow all study-related procedures

Exclusion Criteria:

* Any condition inhibiting MRI study (e.g.Pacemakers or other implantable neurostimulators, ….)
* Subject has any condition, which precludes compliance with study instructions.
* Subject suffers from life threatening conditions
* Anatomical limitations that would prevent successful FMRI study
* Other medical conditions precluding FMRI study - e.g., claustrophobia
* Women gender- due to problematic usage of external urinating device during fMRI study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. 10 Patients with chronic post amputation micturition induced PLP.All subjects must fulfill all of the inclusion criteria and meet none of the exclusion criteria.
  2. 10 Patients with chronic post amputation with PLP and without post amputation micturition induced PLP All subjects must fulfill all of the inclusion criteria and meet none of the exclusion criteria.
  3. 10 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-02-25 (Estimated); Primary Completion 2020-02-02 (Estimated); Study Completion 2020-02-02 (Estimated)

PRIMARY OUTCOMES:
FMRI data analysis | 18 months
  FMRI data analysis signifying, statistically significant uni-spatial voxel activity during micturition, in the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Motti Ratmansky, MD, Principal Investigator — Loewenstein Rehabilitation Hospital
Locations (1):
- Loewenstein Rehabilitation Center, Raanana, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Michels L, Blok BF, Gregorini F, Kurz M, Schurch B, Kessler TM, Kollias S, Mehnert U. Supraspinal Control of Urine Storage and Micturition in Men--An fMRI Study. Cereb Cortex. 2015 Oct;25(10):3369-80. doi: 10.1093/cercor/bhu140. Epub 2014 Jun 26. PMID 24969474
- [Result] Flor H. Phantom-limb pain: characteristics, causes, and treatment. Lancet Neurol. 2002 Jul;1(3):182-9. doi: 10.1016/s1474-4422(02)00074-1. PMID 12849487
- [Result] Shy M, Fung S, Boone TB, Karmonik C, Fletcher SG, Khavari R. Functional magnetic resonance imaging during urodynamic testing identifies brain structures initiating micturition. J Urol. 2014 Oct;192(4):1149-54. doi: 10.1016/j.juro.2014.04.090. Epub 2014 Apr 21. PMID 24769029